CLINICAL TRIAL: NCT05284942
Title: A Trial to Evaluate the Long Term Prognosis in Rosai-Dorfman Disease
Brief Title: Central China Rosai-Dorfman Disease Registry
Acronym: CCR-DDR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, YIKAI YU, Principal Investigator, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: Tongji0509
Record Dates: First submitted 2022-01-18; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Rosai-Dorfman Disease; Langerhans Cell Histiocytosis
MeSH Terms: conditions — Histiocytosis, Sinus; Histiocytosis, Langerhans-Cell | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Mycophenolate mofetil combined with stand of care of oral prednisone 5mg-15mg/day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mycophenolate mofetil (Experimental): Mycophenolate mofetil oral 500mg twice a day from baseline to week 108
  Interventions: Drug: Mycophenolate mofetil combined with oral prednisone

INTERVENTIONS:
Drug: Mycophenolate mofetil combined with oral prednisone — Mycophenolate mofetil oral 500mg twice a day combined with standard of care of oral prednisone 5mg-15mg/day from baseline to week 108

SUMMARY:
This is a research study among patients with Rosai-Dorfman disease.

DETAILED DESCRIPTION:
Rosai-Dorfman disease is a rare disorder characterized by overproduction (proliferation) and accumulation of a specific type of white blood cell (histiocyte) in the lymph nodes of the body (lymphadenopathy), most often those of the neck (cervical lymphadenopathy). In some cases, abnormal accumulation of histiocytes may occur in other areas of the body besides the lymph nodes (extranodal). These areas include the skin, central nervous system, kidney, and digestive tract. The symptoms and physical findings associated with Rosai-Dorfman disease vary depending upon the specific areas of the body that are affected. The disorder predominantly affects mainly adolescents or young adults. The exact cause of Rosa Dorfman disease is unknown. The purpose of this research study is to learn the prevalence , therapies and long term prognosis of Rosa Dorfman disease.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of a histiocytic disorder as determined by a corroborating constellation of histopathology, clinical, and/or radiologic findings. All participants will undergo Standard of Care MRA, CTA or imaging examination.

Exclusion Criteria:

Known intracranial involvement of histiocytosis (including dura, leptomeninges and brain parenchyma) Prior stroke or intracranial hemorrhage Other (non-histiocytic) intracranial neoplasm or neurological disorder deemed by the PI or Co-PI to confound neuroimaging studies (e.g., demyelinating disease) Existing diagnosis of a psychiatric disorder or untreated mood disturbance Existing diagnosis of a neurodegenerative disease, such as Alzheimer's disease Chronic or daily excessive alcohol consumption as determined by the PI. History of chronic use of corticosteroids, defined as continuous treatment for six months or longer at any time in the past History of severe claustrophobia or other contraindications to patient SOC brain MRI Prior intravenous cytarabine or cladribine Other current or prior treatments (e.g., high-dose chemotherapy for a different cancer) deemed by the PI or Co-PI to confound imaging studies or cognitive performance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-10-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Autoimmune bullous disease quality of life (ABQoL) | From baseline to 108 Weeks
  Total ABQoL scores range from 0 to 30 . The ABQoL score is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.

SECONDARY OUTCOMES:
Cumulative Oral Corticosteroid Dose | From 12th, 24th, 36th ,52th and 108 Weeks
  Calculate the Cumulative Oral Corticosteroid Dose

CONTACTS AND LOCATIONS:
Overall Officials: AIHUA DU, M.d, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No